CLINICAL TRIAL: NCT06341361
Title: Optical Coherence Tomography-based Machine Learning for Predicting Fractional Flow Reserve After Coronary Artery Stenting
Brief Title: OCT-based Machine Learning FFR for Predicting Post-PCI FFR
Status: Not yet recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Collaborators: Gangnam Severance Hospital (Other); Severance Hospital (Other)
Responsible Party: Principal Investigator, Jung-Sun Kim, Professor, Yonsei University
Other Study IDs: OCT-FFR
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Tomography, Optical Coherence; Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: OCT-based machine learning FFR — OCT-based machine learning FFR and wire-based FFR

SUMMARY:
This study aims to compare the diagnostic accuracy of the fractional flow reserve (FFR) model derived by machine learning based on optical coherence tomography (OCT) exam after coronary artery stent implantation with the wire-based FFR.

DETAILED DESCRIPTION:
FFR and OCT exam are used for different purposes during percutaneous coronary intervention (PCI). The FFR is a decision-making tool to determine if additional procedures are necessary, while the OCT exam is used to optimize the stent procedure. The use of both tests provides additional information to help perform a excellent procedure, but it is more expensive and time-consuming.

Therefore, an OCT-derived machine learning FFR test may be helpful. Previous studies have demonstrated that OCT-based machine learning FFR before the procedure has shown good diagnostic performance in predicting FFR, irrespective of the coronary territory.

Despite the rapid development of technologies and tools for PCI, a significant number of patients experienced adverse events, such as recurrence of angina and silent ischemia despite angiographically successful PCI. Suboptimal PCI is a well-known independent prognostic factor for major cardiovascular accidents. Therefore, measuring post-PCI FFR immediately after stent implantation is crucial to optimize the procedure outcome and improve the patient's prognosis. Although the importance of measuring post-PCI FFR is gradually emerging, there is currently no model for OCT-based machine learning FFR that predicts FFR after stent insertion. In patients who underwent percutaneous coronary intervention using stents for ischemic heart disease, we will compare the diagnostic accuracy of the fractional flow reserve (FFR) model derived by machine learning based on optical coherence tomography (OCT) exam after coronary artery stent implantation with the wire-based FFR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent stent implantation for ischemic heart disease
2. Patients who underwent both OCT examination and FFR using a pressure wire after PCI

Exclusion Criteria:

1. Poor OCT imaging quality
2. Patients with severe left ventricular dysfunction (<30%)
3. Patients with severe valvular heart disease
4. Patients with a life expectancy of less than 1 year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among patients who underwent PCI for ischemic heart disease, those who underwent both OCT examination and pressure wire-based FFR after coronary artery stenting.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Correlation of OCT-based machine learning FFR compared to wire-based FFR | 4 weeks
  Determining the diagnostic accuracy of CT-FFR values obtained by the new method compared with invasive coronary angiography with fractional flow reserve

SECONDARY OUTCOMES:
Diagnostic performance of OCT-based machine learning FFR compared to wire-based FFR | 4 weeks
  Accuracy, sensitivity, specificity, positive predictive value, negative predictive value
Diagnostic performance of OCT-based machine learning FFR according to the coronary artery (LAD, LCx or RCA) compared to wire-based FFR | 4 weeks
  Accuracy, sensitivity, specificity, positive predictive value, negative predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Sun Kim, MD, PhD, Principal Investigator — Severance Cardiovascular Hospital, Yonsei University College of Medicine

IPD SHARING:
Plan to Share IPD: No